CLINICAL TRIAL: NCT06009276
Title: Associations Between the Microbiome, Skeletal Muscle Perfusion, and Fitness Status
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Professor of Kinesiology, University of Virginia
Other Study IDs: HSR230229
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure, Systolic; Heart Failure, Diastolic; Peripheral Arterial Disease; Overweight and Obesity
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure, Diastolic; Peripheral Arterial Disease; Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart Failure: Patients diagnosed with Heart Failure (HFrEF and HFpEF). Oral microbiome will be analyzed through tongue swabs, saliva samples, and a saliva rinse. Patients will undergo a maximal exercise test, blood draws, and vascular testing. Patients will have the option to participate in a supplementation assessment with concentrated beetroot juice.
- Peripheral Artery Disease: Patients diagnosed with Peripheral Artery Disease (PAD). Oral microbiome will be analyzed through tongue swabs, saliva samples, and a saliva rinse. Patients will undergo a maximal exercise test, blood draws, and vascular testing. Patients will have the option to participate in a supplementation assessment with concentrated beetroot juice.
- Healthy Controls: Individuals that are not diagnosed with cardiovascular disease. Oral microbiome will be analyzed through tongue swabs, saliva samples, and a saliva rinse. Patients will undergo a maximal exercise test, blood draws, and vascular testing. Patients will have the option to participate in a supplementation assessment with concentrated beetroot juice.

SUMMARY:
The purpose of the study is to determine associations between fitness status, bacteria in the mouth, and the blood flow to muscle. This study is trying to find out if fitness status impacts the bacteria that are present in the oral microbiome (environment in the mouth) or the ability of the body to send blood to the skeletal muscle.

Participants will complete all or some of the following:

* A mouth swab to assess the bacteria in their mouths.
* Produce a saliva sample into a tube.
* Cycle on a bike until you reach maximum effort.
* Undergo blood draws
* Wear a 24-hour non-invasive device that monitors blood pressure.
* Drink 70mL (1/3 of a cup) of concentrated beetroot juice once

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in the United States. Nitric oxide (NO) is a gaseous diatomic free-radical and is essential for a plethora of physiological functions involved in cardiometabolic health and CVD risk. NO bioavailability is associated with greater tissue perfusion, mitochondrial function, glucose regulation, and overall reduced CVD risk. The primary source of circulating NO is vascular endothelial nitric oxide synthase.

Unfortunately, the endothelium can be disrupted/damaged via a variety of CVD risk factors such as hypertension, smoking, hyperlipidemia, diabetes, inflammation, and hypercholesteremia. Disruption of the vascular endothelium and loss of bioavailable NO is a preliminary step in the progression of atherosclerosis and CVD. Decreased NO bioavailability and vascular dysfunction have been shown in a variety of clinical conditions including patients heart failure and peripheral artery disease (PAD).

Recently, an exogenous approach to increasing NO bioavailability via oral supplementation of inorganic nitrate (NO3-) has been utilized to increase NO bioavailability in various healthy and clinical populations. Briefly, inorganic NO3- is swallowed, absorbed into the circulation, and sequestered back into the salivary glands. NO3- is then secreted into the oral cavity, where bacteria containing nitrate reductase enzymes convert NO3- to nitrite (NO2-), which is again swallowed and absorbed into the circulation. NO2- in the plasma is then easily reduced to NO via non-enzymatic reactions.

This study aims to better elucidate the relationship between the oral microbiome abundance and diversity and NO3- to NO2- to NO conversion across a variety of subject populations ranging from healthy subjects to those with risk factors for CVD and people with diagnosed CVD. We also aim to examine the relationship between oral microbiome NO3- reduction and impaired skeletal muscle perfusion and exercise capacity as NO bioavailability plays a large role in these physiological processes.

The results of this study may allow us to better understand how novel interventions to modify the oral microbiome may improve cardiometabolic health and physical function in individuals with CVD and outline potential new therapeutic approaches.

The primary objective of this preliminary study is to compare the abundance and diversity of oral NO3- reducing bacteria in a variety of subjects with varying cardiometabolic health status and their ability to convert oral inorganic nitrate to nitrite measured in the saliva and plasma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Subjects may be of either sex with age 18 years.

Exclusion Criteria:

* Oral antibiotic use within previous four weeks
* Oral disease or poor oral health as determined by the Oral Health Questionnaire
* Using an antibacterial mouthwash or a mouthwash containing chlorhexidine and unwilling to discontinue use
* Tobacco smokers
* Pregnant or lactating females
* Hypersensitivity to any ultrasound contrast agent
* Inability to perform exercise
* Unable to communicate effectively in English to the study team.
* Diagnosis of chronic renal failure (GFR < 60 ml/min/1.73m)
* Subjects taking nitroglycerine (or inorganic nitrates), PDE-5 inhibitors (ex: Cialis, Viagra), and xanthine oxidase inhibitors (ex: Allopurinol).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population will include healthy individuals over the age of 18 years of either sex, or individuals with cardiovascular disease (heart failure, peripheral artery disease).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Oral Nitrate Reducing Capacity | Baseline, 4-weeks, 12-weeks, 6-months
  Assessment of the oral microbiome's ability to reduce nitrate to nitrite. This will be measured through a swab on the dorsal surface of the tongue, an unstimulated saliva sample, and a rinse of a standard nitrate solution.

SECONDARY OUTCOMES:
Aerobic Capacity | Baseline, 4-weeks, 12-weeks, 6-months
  Peak aerobic capacity (VO2peak) will be assessed using a symptom-limited graded exercise test on a cycle ergometer.

OTHER OUTCOMES:
Peripheral and Central Blood Pressures | Baseline, 4-weeks, 12-weeks, 6-months
  Brachial artery blood pressures will be obtained using a standard sphygmomanometer. Aortic blood pressures will be obtained using applanation tonometry (SphygmoCor version 8.0, AtCor Medical).
24-hour ambulatory blood pressure | Baseline, 4-weeks, 12-weeks, 6-months
  Blood pressure will be monitored using a standard ambulatory brachial artery blood pressure cuff (SunTech Oscar 2, SunTech Medical). Blood pressure measurements are programmed to be taken every 30-minutes during the day and every hour at night. This allows for monitoring of nighttime blood pressure changes and variations throughout the day.
Flow-Mediated Dilation | Baseline, 4-weeks, 12-weeks, 6-months
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The arteries will be imaged using a high-resolution 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 3 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle.
Serum Glucose | Baseline, 4-weeks, 12-weeks, 6-months
  A blood sample will be obtained to measure serum glucose.
Insulin | Baseline, 4-weeks, 12-weeks, 6-months
  A blood sample will be obtained to measure insulin.
Lipids | Baseline, 4-weeks, 12-weeks, 6-months
  A blood sample will be obtained to measure lipids.
Hemoglobin | Baseline, 4-weeks, 12-weeks, 6-months
  A blood sample will be obtained to measure hemoglobin.
Hematocrit | Baseline, 4-weeks, 12-weeks, 6-months
  A blood sample will be obtained to measure hematocrit.
Plasma Nitrate | Baseline, 4-weeks, 12-weeks, 6-months
  A fasting blood draw will be taken. Following the blood draw, the participant will take one dose of Beetroot juice. The participant will then return to the lab three hours later for a second blood draw to assess level of nitrate in the plasma.
Plasma Nitrite | Baseline, 4-weeks, 12-weeks, 6-months
  A fasting blood draw will be taken. Following the blood draw, the participant will take one dose of Beetroot juice. The participant will then return to the lab three hours later for a second blood draw to assess level of nitrite in the plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Allen, PhD, Principal Investigator — University of Virginia
Locations (1):
- UVA Student Health and Wellness Building, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No